CLINICAL TRIAL: NCT06281262
Title: The Role of Selected Immunological Indicators and Microbiota in Patients Experiencing Premature Birth and Preeclampsia
Brief Title: Selected Immunological Indicators and Microbiota in Patients With Premature Birth and Preeclampsia
Acronym: PRIME
Status: Recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Collaborators: Charles University, Czech Republic (Other); Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Responsible Party: Principal Investigator, Zdenek Lastuvka, Principal investigator, MD, General University Hospital, Prague
Other Study IDs: GIP-23-L-04-223
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Preeclampsia
Keywords: Preterm labor; Regulatory T cells; Early pregnancy; Immunology; Maternal-fetal interface
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Flow cytometry includes a live/dead discriminator dye and markers for identification of major T cells and NK cell lineages as well as functional markers. Data will be analyzed using a hybrid approach combining manual gating in FlowJo and unsupervised clustering using the GQT-SOM dimensionality reduction algorithm collaboratively developed between IHBT and IOCB. Flow cytometry will be used to test Treg suppressive function by measuring the suppression of target cell proliferation in carboxyfluorescein succinimidyl ester (CFSE) dilution assay, coculturing CFSE-stained target cells (CBMC or CD4+CD25-). Bacterial DNA will be isolated from oral, vaginal, rectal swabs and piece of placenta for determination of bacterial species according to bacterial 16S rRNA. We will utilise Illumina MiSeq platform, where specific region of 16S rRNA (region V4) will be sequenced and followed by sophisticated analysis (LEfSe). Sequencing will be outsourced to Laboratory of Environmental Microbiology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Singletone pregnancy, gestational age 9+0 - 12+0, history of preeclampsia (PE) or spontaneous preterm birth (PTL = preterm labour) or pPROM (preterm premature rupture of membranes).
  Interventions: Diagnostic Test: Peripheral blood collection; Diagnostic Test: Swab sample collection

INTERVENTIONS:
Diagnostic Test: Peripheral blood collection — The phenotypic characteristics of leukocytes will be compared between the groups to identify immunological markers of women at risk of preterm delivery.
  Samples from the controls will be taken to define a baseline for the measured leukocyte populations.
Diagnostic Test: Swab sample collection — Oral, vaginal and rectal swabs will be collected and stored for analysis of microbiota at the time of inclusion. At birth, oral, vaginal and rectal swabs and part of the placenta (placental tissue) will be collected for further analysis.

SUMMARY:
The goal is to demonstrate the relationship of the circulating pool of T-regulatory lymphocytes in the mother's peripheral blood with populations in the placentas and to compare with controls, what is the difference in the expression of individual regulatory molecules of T-regulatory lymphocytes according to new paradigms. The proportional and functional characteristics of T-regulatory lymphocytes will be correlated with the composition of the intestinal and vaginal microbiota.

DETAILED DESCRIPTION:
OBJECTIVES

The primary objective of this project is to determine the differences between the circulating pool of regulatory Treg subpopulation proportions and the placental populations in patients with preterm birth and preeclampsia. Pilot study was conducted for the primary objective. Another objective is to evaluate the effect of microbiota on the regulation of Treg cells, especially in relation to mechanisms of preterm birth and preeclampsia. With growing knowledge of the role of microbiota, it is considered that the maternal microbiota could significantly influence setting of immunoregulatory responses even prenatally. Since Treg play a key role in regulating the immunological balance and are indispensable for induction and maintenance of peripheral tolerance, the investigators hypothesise that abnormalities in function of this population are important factors in increasing the risk of gestational pathologies (preterm birth and preeclampsia). Such dysregulation is most likely accompanied by disruption of the physiological Treg epigenetic profile which is in turn influenced by aberrant microbiota composition. Better understanding of these processes and identification of positively or negatively participating bacterial species could enable more reliable prediction of risk-pregnancy and allow for modulation of microbiota to be applied preventively.

Premature birth is defined as pregnancy termination before the end of the gestational week 37. It plays a role in 10% of all pregnancies including spontaneous or medically induced labours. The efforts to postpone premature labour are continuously developed to minimise the consequences such as low birth weight and other risk events. Preeclampsia is a serious blood pressure condition that develops during pregnancy. People with preeclampsia often have high blood pressure (hypertension) and high levels of protein in their urine (proteinuria). It plays role in 5% of all pregnancies. Preeclampsia typically develops after the 20th week of pregnancy. It can also affect other organs in the body and be dangerous for both the mother and her unborn child. Therefore, a great number of scientific studies are now focused on the early prediction of premature labour and preeclampsia and on finding a specific parameter to estimate female patients at premature labour and preeclampsia risk.

HYPOTHESIS AND AIMS

Hypothesis 1: Disbalance between tolerogenic T cell subsets (Treg, Th2, Th9 and Th22) and proinflammatory subsets (Th1 and Th17) is a sign of premature birth or preeclampsia.

Specific aim 1: Determine the differences between the circulating and the placental T cell subpopulations in patients with preterm birth and preeclampsia. Previously published analyses of Trees and their phenotypic properties give inconclusive or even contradictory results. For this reason, the investigators propose a more in depth approach combining deep immunophenotyping capable of identifying effector T cell, Treg and NK cell subsets and their qualitative phenotype together with assessment of functional capabilities of Tregs.

Hypothesis 2: Certain bacterial species of microbiota can be identified to modulate epigenetic maintenance of Treg phenotype.

Specific aim 2: Determine the influence of microbiota on the Treg regulation. Exposure to microbiota is one of the most important environmental factors introduced in the perinatal period. The capability of certain probiotic bacterial species to promote immunological tolerance, restrain inflammation and unwanted reactivity is being established in the context of intestinal health. Both bacteria and their metabolic products are known to shape the immune system. By influencing the epigenetic programming they modulate phenotype and function of a variety of immune cells including Tregs. The investigators hypothesise that beneficial bacterial species can be identified to promote appropriate epigenetic maintenance of Treg phenotype, function and stability, and thus support Treg tolerogenic role. On the contrary, certain bacterial species will contribute to Treg epigenetic dysregulation and introduce a more pro-inflammatory environment with functionally deficient Treg cells. To test this hypothesis, the investigators will characterise microbial composition of material collected from the mother by oral, rectal and vaginal swabs during pregnancy and at the time of birth.

CHARACTERISATION OF EXPECTED RESULTS

The main outcome of the project will be to improve the understanding of the regulatory processes taking part in the immune balance in preterm birth and preeclampsia. Special attention will be given to the dynamics and functional characteristics of Treg and their subpopulations, considering the role of maternal microbiota. The obtained results will be presented on both national and international congresses and symposia and also published in international impacted journals.

ELIGIBILITY:
Inclusion Criteria:

* singletone pregnancy
* gestational age 9+0 - 12+0
* history of preeclampsia (PE)
* history of spontaneous preterm birth (PTL = preterm labour)
* history of pPROM (preterm premature rupture of membranes).

Exclusion Criteria:

* uterine malformations
* gestational age out of 9+0 - 12+0
* age out of 19-40

Ages: 19 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in selected T cell subpopulations in the first trimester associated with subsequent spontaneous preterm birth | 3 years
  The phenotypic characteristics of leukocytes will be compared between the two groups of pregnant women to identify immunological markers of preterm delivery. Peripheral blood from age-matched healthy nonpregnant women (N=20) will also be collected to define a baseline for the measured leukocyte populations. Furthermore, the composition of placenta infiltrating lymphocytes will be compared between groups and following delivery.
Changes in selected T cell subpopulations in the first trimester associated with subsequent pre-eclampsia | 3 years
  The phenotypic characteristics of leukocytes will be compared between the two groups of pregnant women to identify immunological markers of pre-eclampsia. Peripheral blood from age-matched healthy nonpregnant women (N=20) will also be collected to define a baseline for the measured leukocyte populations. Furthermore, the composition of placenta infiltrating lymphocytes will be compared between groups and following delivery.

SECONDARY OUTCOMES:
Association of maternal microbiota and maternal T regulatory cell populations. | 3 years
  At birth, oral, vaginal and rectal swabs and part of the placenta (placental tissue) will be collected for analysis. Microbial composition of the swabs will be analysed using 16S rRNA sequencing analysis of microbiota and put in context with the T-cell regulatory population of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Zdeněk Laštůvka, MD, PhD, Principal Investigator — General University Hospital, Prague
Locations (1):
- Department of Gynaecology, Obstetrics and Neonatology of the First Faculty of Medicine of the Charles University and General University Hospital in Prague, Prague, Czechia

REFERENCES:
- [Background] Perin J, Mulick A, Yeung D, Villavicencio F, Lopez G, Strong KL, Prieto-Merino D, Cousens S, Black RE, Liu L. Global, regional, and national causes of under-5 mortality in 2000-19: an updated systematic analysis with implications for the Sustainable Development Goals. Lancet Child Adolesc Health. 2022 Feb;6(2):106-115. doi: 10.1016/S2352-4642(21)00311-4. Epub 2021 Nov 17. PMID 34800370
- [Background] Ohuma EO, Moller AB, Bradley E, Chakwera S, Hussain-Alkhateeb L, Lewin A, Okwaraji YB, Mahanani WR, Johansson EW, Lavin T, Fernandez DE, Dominguez GG, de Costa A, Cresswell JA, Krasevec J, Lawn JE, Blencowe H, Requejo J, Moran AC. National, regional, and global estimates of preterm birth in 2020, with trends from 2010: a systematic analysis. Lancet. 2023 Oct 7;402(10409):1261-1271. doi: 10.1016/S0140-6736(23)00878-4. PMID 37805217
- [Background] Manuck TA. Racial and ethnic differences in preterm birth: A complex, multifactorial problem. Semin Perinatol. 2017 Dec;41(8):511-518. doi: 10.1053/j.semperi.2017.08.010. Epub 2017 Sep 21. PMID 28941962
- [Background] Chawanpaiboon S, Vogel JP, Moller AB, Lumbiganon P, Petzold M, Hogan D, Landoulsi S, Jampathong N, Kongwattanakul K, Laopaiboon M, Lewis C, Rattanakanokchai S, Teng DN, Thinkhamrop J, Watananirun K, Zhang J, Zhou W, Gulmezoglu AM. Global, regional, and national estimates of levels of preterm birth in 2014: a systematic review and modelling analysis. Lancet Glob Health. 2019 Jan;7(1):e37-e46. doi: 10.1016/S2214-109X(18)30451-0. Epub 2018 Oct 30. PMID 30389451
- [Background] Ream MA, Lehwald L. Neurologic Consequences of Preterm Birth. Curr Neurol Neurosci Rep. 2018 Jun 16;18(8):48. doi: 10.1007/s11910-018-0862-2. PMID 29907917
- [Background] Green ES, Arck PC. Pathogenesis of preterm birth: bidirectional inflammation in mother and fetus. Semin Immunopathol. 2020 Aug;42(4):413-429. doi: 10.1007/s00281-020-00807-y. Epub 2020 Sep 7. PMID 32894326
- [Background] Gomez-Lopez N, Arenas-Hernandez M, Romero R, Miller D, Garcia-Flores V, Leng Y, Xu Y, Galaz J, Hassan SS, Hsu CD, Tse H, Sanchez-Torres C, Done B, Tarca AL. Regulatory T Cells Play a Role in a Subset of Idiopathic Preterm Labor/Birth and Adverse Neonatal Outcomes. Cell Rep. 2020 Jul 7;32(1):107874. doi: 10.1016/j.celrep.2020.107874. PMID 32640239
- [Background] Robertson SA, Care AS, Moldenhauer LM. Regulatory T cells in embryo implantation and the immune response to pregnancy. J Clin Invest. 2018 Oct 1;128(10):4224-4235. doi: 10.1172/JCI122182. Epub 2018 Oct 1. PMID 30272581
- [Background] Xue L, Gyles SL, Wettey FR, Gazi L, Townsend E, Hunter MG, Pettipher R. Prostaglandin D2 causes preferential induction of proinflammatory Th2 cytokine production through an action on chemoattractant receptor-like molecule expressed on Th2 cells. J Immunol. 2005 Nov 15;175(10):6531-6. doi: 10.4049/jimmunol.175.10.6531. PMID 16272307
- [Background] Tsuda S, Zhang X, Hamana H, Shima T, Ushijima A, Tsuda K, Muraguchi A, Kishi H, Saito S. Clonally Expanded Decidual Effector Regulatory T Cells Increase in Late Gestation of Normal Pregnancy, but Not in Preeclampsia, in Humans. Front Immunol. 2018 Aug 24;9:1934. doi: 10.3389/fimmu.2018.01934. eCollection 2018. PMID 30197648
- [Background] Rowe JH, Ertelt JM, Xin L, Way SS. Pregnancy imprints regulatory memory that sustains anergy to fetal antigen. Nature. 2012 Oct 4;490(7418):102-6. doi: 10.1038/nature11462. Epub 2012 Sep 26. PMID 23023128
- [Background] Schober L, Radnai D, Schmitt E, Mahnke K, Sohn C, Steinborn A. Term and preterm labor: decreased suppressive activity and changes in composition of the regulatory T-cell pool. Immunol Cell Biol. 2012 Nov;90(10):935-44. doi: 10.1038/icb.2012.33. Epub 2012 Jul 3. PMID 22751216
- [Background] Tilburgs T, Roelen DL, van der Mast BJ, de Groot-Swings GM, Kleijburg C, Scherjon SA, Claas FH. Evidence for a selective migration of fetus-specific CD4+CD25bright regulatory T cells from the peripheral blood to the decidua in human pregnancy. J Immunol. 2008 Apr 15;180(8):5737-45. doi: 10.4049/jimmunol.180.8.5737. PMID 18390759
- [Background] Krop J, Heidt S, Claas FHJ, Eikmans M. Regulatory T Cells in Pregnancy: It Is Not All About FoxP3. Front Immunol. 2020 Jun 23;11:1182. doi: 10.3389/fimmu.2020.01182. eCollection 2020. PMID 32655556
- [Background] Green S, Politis M, Rallis KS, Saenz de Villaverde Cortabarria A, Efthymiou A, Mureanu N, Dalrymple KV, Scotta C, Lombardi G, Tribe RM, Nicolaides KH, Shangaris P. Regulatory T Cells in Pregnancy Adverse Outcomes: A Systematic Review and Meta-Analysis. Front Immunol. 2021 Oct 29;12:737862. doi: 10.3389/fimmu.2021.737862. eCollection 2021. PMID 34777347
- [Background] Tsuda S, Nakashima A, Shima T, Saito S. New Paradigm in the Role of Regulatory T Cells During Pregnancy. Front Immunol. 2019 Mar 26;10:573. doi: 10.3389/fimmu.2019.00573. eCollection 2019. PMID 30972068
- [Background] Rudensky AY. Regulatory T cells and Foxp3. Immunol Rev. 2011 May;241(1):260-8. doi: 10.1111/j.1600-065X.2011.01018.x. PMID 21488902
- [Background] Yadav M, Stephan S, Bluestone JA. Peripherally induced tregs - role in immune homeostasis and autoimmunity. Front Immunol. 2013 Aug 7;4:232. doi: 10.3389/fimmu.2013.00232. eCollection 2013. PMID 23966994
- [Background] Elkord E. Helios Should Not Be Cited as a Marker of Human Thymus-Derived Tregs. Commentary: Helios(+) and Helios(-) Cells Coexist within the Natural FOXP3(+) T Regulatory Cell Subset in Humans. Front Immunol. 2016 Jul 8;7:276. doi: 10.3389/fimmu.2016.00276. eCollection 2016. No abstract available. PMID 27456241
- [Background] Kim HJ, Barnitz RA, Kreslavsky T, Brown FD, Moffett H, Lemieux ME, Kaygusuz Y, Meissner T, Holderried TA, Chan S, Kastner P, Haining WN, Cantor H. Stable inhibitory activity of regulatory T cells requires the transcription factor Helios. Science. 2015 Oct 16;350(6258):334-9. doi: 10.1126/science.aad0616. PMID 26472910
- [Background] Yu WQ, Ji NF, Gu CJ, Wang YL, Huang M, Zhang MS. Coexpression of Helios in Foxp3+ Regulatory T Cells and Its Role in Human Disease. Dis Markers. 2021 Jun 22;2021:5574472. doi: 10.1155/2021/5574472. eCollection 2021. PMID 34257746
- [Background] Shevyrev D, Tereshchenko V. Treg Heterogeneity, Function, and Homeostasis. Front Immunol. 2020 Jan 14;10:3100. doi: 10.3389/fimmu.2019.03100. eCollection 2019. PMID 31993063
- [Background] Zhao H, Bo C, Kang Y, Li H. What Else Can CD39 Tell Us? Front Immunol. 2017 Jun 22;8:727. doi: 10.3389/fimmu.2017.00727. eCollection 2017. PMID 28690614
- [Background] Svensson-Arvelund J, Mehta RB, Lindau R, Mirrasekhian E, Rodriguez-Martinez H, Berg G, Lash GE, Jenmalm MC, Ernerudh J. The human fetal placenta promotes tolerance against the semiallogeneic fetus by inducing regulatory T cells and homeostatic M2 macrophages. J Immunol. 2015 Feb 15;194(4):1534-44. doi: 10.4049/jimmunol.1401536. Epub 2015 Jan 5. PMID 25560409
- [Background] Wang S, Zhu X, Xu Y, Zhang D, Li Y, Tao Y, Piao H, Li D, Du M. Programmed cell death-1 (PD-1) and T-cell immunoglobulin mucin-3 (Tim-3) regulate CD4+ T cells to induce Type 2 helper T cell (Th2) bias at the maternal-fetal interface. Hum Reprod. 2016 Apr;31(4):700-11. doi: 10.1093/humrep/dew019. Epub 2016 Feb 16. PMID 26908841
- [Background] Wang W, Sung N, Gilman-Sachs A, Kwak-Kim J. T Helper (Th) Cell Profiles in Pregnancy and Recurrent Pregnancy Losses: Th1/Th2/Th9/Th17/Th22/Tfh Cells. Front Immunol. 2020 Aug 18;11:2025. doi: 10.3389/fimmu.2020.02025. eCollection 2020. PMID 32973809
- [Background] Travis OK, White D, Pierce WA, Ge Y, Stubbs CY, Spradley FT, Williams JM, Cornelius DC. Chronic infusion of interleukin-17 promotes hypertension, activation of cytolytic natural killer cells, and vascular dysfunction in pregnant rats. Physiol Rep. 2019 Apr;7(7):e14038. doi: 10.14814/phy2.14038. PMID 30963715
- [Background] Wang WJ, Hao CF, Yi-Lin, Yin GJ, Bao SH, Qiu LH, Lin QD. Increased prevalence of T helper 17 (Th17) cells in peripheral blood and decidua in unexplained recurrent spontaneous abortion patients. J Reprod Immunol. 2010 Mar;84(2):164-70. doi: 10.1016/j.jri.2009.12.003. Epub 2010 Jan 27. PMID 20106535
- [Background] van der Zwan A, Bi K, Norwitz ER, Crespo AC, Claas FHJ, Strominger JL, Tilburgs T. Mixed signature of activation and dysfunction allows human decidual CD8+ T cells to provide both tolerance and immunity. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):385-390. doi: 10.1073/pnas.1713957115. Epub 2017 Dec 19. PMID 29259116
- [Background] Jabrane-Ferrat N. Features of Human Decidual NK Cells in Healthy Pregnancy and During Viral Infection. Front Immunol. 2019 Jun 28;10:1397. doi: 10.3389/fimmu.2019.01397. eCollection 2019. PMID 31379803
- [Background] Moffett-King A. Natural killer cells and pregnancy. Nat Rev Immunol. 2002 Sep;2(9):656-63. doi: 10.1038/nri886. PMID 12209134
- [Background] Thomsen SF. Epidemiology and natural history of atopic diseases. Eur Clin Respir J. 2015 Mar 24;2. doi: 10.3402/ecrj.v2.24642. eCollection 2015. PMID 26557262
- [Background] Hagihara Y, Yoshimatsu Y, Mikami Y, Takada Y, Mizuno S, Kanai T. Epigenetic regulation of T helper cells and intestinal pathogenicity. Semin Immunopathol. 2019 May;41(3):379-399. doi: 10.1007/s00281-019-00732-9. Epub 2019 Mar 19. PMID 30891628
- [Background] Berni Canani R, Paparo L, Nocerino R, Di Scala C, Della Gatta G, Maddalena Y, Buono A, Bruno C, Voto L, Ercolini D. Gut Microbiome as Target for Innovative Strategies Against Food Allergy. Front Immunol. 2019 Feb 15;10:191. doi: 10.3389/fimmu.2019.00191. eCollection 2019. PMID 30828329
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Nakashima A, Ito M, Shima T, Bac ND, Hidaka T, Saito S. Accumulation of IL-17-positive cells in decidua of inevitable abortion cases. Am J Reprod Immunol. 2010 Jul 1;64(1):4-11. doi: 10.1111/j.1600-0897.2010.00812.x. Epub 2010 Mar 4. PMID 20219063
- [Background] Vanikova S, Koladiya A, Musil J. OMIP-080: 29-Color flow cytometry panel for comprehensive evaluation of NK and T cells reconstitution after hematopoietic stem cells transplantation. Cytometry A. 2022 Jan;101(1):21-26. doi: 10.1002/cyto.a.24510. Epub 2021 Oct 24. PMID 34693626
- [Background] Kratochvil M, Koladiya A, Vondrasek J. Generalized EmbedSOM on quadtree-structured self-organizing maps. F1000Res. 2019 Dec 18;8:2120. doi: 10.12688/f1000research.21642.2. eCollection 2019. PMID 32518625